CLINICAL TRIAL: NCT03646825
Title: Observation Study of the Effect of Use of Natural Antioxidant Supplement on Sperm DNA Fragmentation
Brief Title: Effect of Natural Antioxidant Supplement on Sperm DNA Fragmentation
Status: Terminated | Type: Observational
Why Stopped: Completed study with fewer participants than expected
Sponsor: Colorado Center for Reproductive Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 20170532
Record Dates: First submitted 2018-08-23; First posted 2018-08-24 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Observe Effect of Antioxidant on Sperm DNA Fragmention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment group: Male patients exposed to antioxidant for 12 weeks
  Interventions: Dietary Supplement: Natural Antioxidant supplement

INTERVENTIONS:
Dietary Supplement: Natural Antioxidant supplement — 1 capsule orally three times a day for 12 weeks

SUMMARY:
Observational study to see the effect of use of natural Antioxidant supplement on sperm DNA fragmentation. Subjects will take the natural antioxidant for 3 months prior to repeat testing.

DETAILED DESCRIPTION:
Male patients will be recruited based on having a high DNA fragmentation (chromatin >16) no other severe male factor infertility (>5million/ml, count, > 10%motility and >1% morphology) and sufficient ejaculate sperm for ICSI (no surgically removed sperm or history of vasectomy reversal). Patients will be provided the natural antioxidant supplementation by the sponsor. Patients will take 1 capsule orally 3 times a day for a full 12 weeks. Sperm DNA structure will be re-assessed after completion of 12 weeks of antioxidant to compare to baseline sperm DNA structure collected prior to starting regimen of supplement daily

ELIGIBILITY:
Inclusion Criteria:

-Sperm Chromatin >16%, sufficient ejaculate sperm for ICSI

Exclusion Criteria:

* Severe male factor infertility

Ages: 18 Years to 55 Years | Sex: Male
Age Groups: Adult
Study Population: Male patients pursuing IVF for treatment of infertility
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Sperm DNA fragmentation | 12 weeks
  Direct comparison of sperm DNA fragmentation pre and post natural antioxidant exposure

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Makloski, Study Chair — Study Coordinator
Locations (1):
- Colorado Center for Reproductive Medicine, Lone Tree, Colorado, United States

IPD SHARING:
Plan to Share IPD: No